CLINICAL TRIAL: NCT07308483
Title: Ketogenic Approach to Restore Muscle in Older Patients With Community-Acquired Pneumonia - KARMA-P Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Robert T Mankowski, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300015253; 1R21AG098466-01 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2025-11-17; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia
Keywords: ketogenic feeding; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketogenic feeding (Active Comparator): The ketogenic feeding will have a macronutrient composition of approximately 10% energy from carbohydrates, 25% energy from protein, and 65% energy from fat.
  Interventions: Behavioral: Ketogenic feeding
- Standard feeding (Placebo Comparator): The standard, control diet will be compatible with the USDA guidelines. It will consist of approximately 60% carbohydrate, 20% protein, 20% fat. Participants will be given low-fat foods, whole-grain foods, fruits, and vegetables.
  Interventions: Behavioral: Standard feeding

INTERVENTIONS:
Behavioral: Ketogenic feeding — The ketogenic feeding will have a macronutrient composition of approximately 10% energy from carbohydrates, 25% energy from protein, and 65% energy from fat. No food group will be excluded in this diet prescription; however, the diet will emphasize low-glycemic sources of carbohydrate, and include mainly whole foods such as non-starchy vegetables with minimal highly processed grain products and added sugar. Protein foods will include meat, poultry, fish, eggs, and whey protein supplements, if necessary. Fat-containing foods will include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; avocados; and the fat found in meat. A number of full-fat dairy products will be included. Saturated fat will be limited to 10% of total fat intake. Patients will obtain the majority of their fat intake from poly- and mono-unsaturated fatty acids at a 4:1 ratio.
  Arms: ketogenic feeding
Behavioral: Standard feeding — The standard, control diet will be compatible with the USDA guidelines. It will consist of approximately 60% carbohydrate, 20% protein, 20% fat. Participants will be given low-fat foods, whole-grain foods, fruits, and vegetables. The meal plans will minimize cholesterol, high-fat foods, high-cholesterol foods, processed starches, and added sugar, and will provide <2300 mg/day sodium. Saturated fat will be limited to 10% of total fat intake, and all dairy products will be fat-free (or low fat). Participants will obtain the majority of their fat intake from poly- and mono-unsaturated fatty acids at a 4:1 ratio matched to the ketogenic feeding group; however, total grams will be lower.
  Arms: Standard feeding

SUMMARY:
The purpose of the study is to see if a ketogenic diet compared to a standard diet is better to maintain muscle function and health in hospital admitted pneumonia patients.

DETAILED DESCRIPTION:
Bacterial community-acquired pneumonia (CAP) is a leading cause of hospitalization and mortality in older adults, often resulting in significant muscle wasting, systemic inflammation, and microbiome dysbiosis. Muscle loss, driven by bedrest, acute illness, and antibiotic-induced dysbiosis, all contribute to prolonged hospital stay, delayed recovery, and long-term physical decline. Current interventions such as physical rehabilitation and increased protein intake are largely ineffective in mitigating the acute illness-induced muscle wasting due to metabolic dysfunction such as impaired glucose control. Preliminary evidence suggests that ketogenic enteral feeding is safe, reduces inflammation, stabilizes metabolism and preserves functional outcomes in hospitalized patients. Because most of older hospitalized CAP patients are able to ingest food orally, our study aims to test the safety, feasibility and determine effect sizes for preliminary evidence of a 10-day oral ketogenic diet (low carbohydrate, high fat) in older CAP patients.

The investigators will conduct a double-blinded pilot randomized clinical trial in 30 hospitalized older adults (>55 years) with bacterial CAP, randomizing participants to a ketogenic feeding (n=15) or standard hospital feeding (n=15). Muscle mass will be assessed using ultrasound, inflammatory and metabolic biomarkers from blood, and microbiome composition from oral and skin swabs collected at baseline, 10-Day post-intervention, and 1-month post-intervention follow-up. Handgrip strength will be collected at baseline and 10-day follow-up. Physical activity measures (accelerometry) will be measured for 7 days after the 10-day and 1-month follow-up visits. Physical function (short physical performance battery), handgrip strength, and activity levels (accelerometry) will be measured at 1-month follow-up. Daily blood ketone level measurements will guide feeding adjustments to maintain ketosis, and dietary habits will be assessed weekly post-intervention until 1-month follow-up. Meals for the 10-day intervention will be prepared in a metabolic kitchen by a clinical nutritionist.

If successful, this study will provide evidence for oral ketogenic feeding as an innovative intervention to prevent muscle wasting and functional decline, supporting a future phase IIb clinical trial targeting middle-aged and older adults hospitalized with CAP.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years and older
* Bacterial community-acquired pneumonia
* Expected at least 10-day stay in the hospital
* Ability to ingest food orally
* Willingness to be randomized to either treatment group
* Willingness to participate in all study procedures

Exclusion Criteria:

* Failure to provide informed consent
* Moribund
* Vegetarian/vegan
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Diagnosed dementia
* Hip fracture, hip or knee replacement, or spinal surgery within past 4 months
* Simultaneous participation in another intervention trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | At baseline, at 10-day of feeding, and at 1 month follow-up
  Number of adverse events collected using a standardized adverse event reporting form (Unit: Count of events).
Adherence to the Intervention | From baseline to 1 month follow-up
  Percentage of prescribed intervention sessions completed, assessed through adherence logs and system usage records (Unit: %)

SECONDARY OUTCOMES:
Handgrip strength | At baseline, 10-Day post-intervention, and 1-month post-intervention follow-up
  Participants will be asked to squeeze a metal handle of a dynamometer device as hard as possible at 2 trials, which will be averaged (Unit: Kilograms).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided